CLINICAL TRIAL: NCT01684540
Title: Non-interventional Study: Application of Ectoin® Rhinitis Nasal Spray in Patients With Acute Rhinosinusitis
Brief Title: Application of Ectoin® Rhinitis Nasal Spray in Patients With Acute Rhinosinusitis
Acronym: SNS01
Status: Completed | Type: Observational
Sponsor: Bitop AG (Industry)
Responsible Party: Sponsor
Other Study IDs: PPL-047; NIS SNS01
Record Dates: First submitted 2012-09-11; First posted 2012-09-13 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Sinusitis
Keywords: sinusitis, rhinosinusitis, ectoin, ectoine, bitop, SNS, SNS01
MeSH Terms: conditions — Sinusitis; Rhinosinusitis | interventions — Equipment and Supplies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Medical Device, Drug-like — Ectoin Rhinitis Nasal Spray
Drug: Sinupret forte

SUMMARY:
This is a comparative, open label, parallel group, non interventional study to further demonstrate the effectiveness and tolerability of Ectoin® Rhinitis Nasal Spray. In addition the effectiveness and safety shall be compared to a Sinupret forte. The patient applies Ectoin® Rhinitis Nasal Spray or takes Sinupret forte according to the instructions for use. The observation takes place over a period of 14 days. Response to treatment is recorded at day 7 and day 14 by the physician and in daily by the patient in a dairy.

ELIGIBILITY:
Inclusion Criteria:

* Female or male individuals ≥ 18 years
* Patients with acute Rhinosinusitis which are treated with Ectoin® Rhinitis Nasal Spray or Sinupret forte during the observational period

Exclusion Criteria:

* Contra indications according to the label

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2012-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Changes in the symptoms of acute Rhinosinusitis assessed by the EPOS- Sinusitis-Symptom-Score | day 1, day 7, day 14

SECONDARY OUTCOMES:
Quality of Life questionnaire (Rhino QoL) | day 1, day 7, day 14
Rhinoscopy | day 1, day 7, day 14
Patient's and physician's judgment of efficacy | day 7, day 14

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Mösges, Prof., Study Director — Institut für Med. Informatik, Statistik und Epidemiologie
Locations (6):
- Germany (6):
  - Dr. med. Georg Krueckels, Aachen
  - Dr. med. Martin Sondermann, Aachen
  - Dr. med. Norbert Pasch, Aachen
  - Peter Hinterkausen, Cologne
  - Taufik Shahab, Cologne
  - Dr. med. Wilhelm Schuetz, Jülich

REFERENCES:
- [Derived] Eichel A, Wittig J, Shah-Hosseini K, Mosges R. A prospective, controlled study of SNS01 (ectoine nasal spray) compared to BNO-101 (phytotherapeutic dragees) in patients with acute rhinosinusitis. Curr Med Res Opin. 2013 Jul;29(7):739-46. doi: 10.1185/03007995.2013.800474. Epub 2013 May 14. PMID 23621514